CLINICAL TRIAL: NCT07322432
Title: The CONQUER Trial: Cessation Of Nicotine, QUitting With E-cigarette Reduction - A Single-Arm, Open-Label Clinical Trial to Assess the Efficacy of VapeAway in Promoting Vaping Cessation Compared to Historical Rates of Vaping Cessation
Brief Title: The CONQUER Trial - Cessation Of Nicotine, QUitting With E-cigarette Reduction
Acronym: CONQUER
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: VapeAway (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2025-VPA-001
Record Dates: First submitted 2026-01-01; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Addiction Nicotine
Keywords: Vaping; Vaping Addiction; Vaping Cessation; Vape
MeSH Terms: conditions — Tobacco Use Disorder; Vaping

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Intervention Arm (Experimental): Participants with a vaping addiction that use the VapeAway system to help vaping cessation
  Interventions: Device: VapeAway filter system

INTERVENTIONS:
Device: VapeAway filter system — A multi-component, drug-free program for vaping cessation. The system integrates three core elements: nicotine tapering filters, fix bar behavioral substitution tool, digital support system.

SUMMARY:
This clinical trial evaluates the VapeAway system, a novel, multi-modal intervention designed to address the multifaceted nature of vaping addiction. VapeAway combines progressive nicotine tapering via proprietary filters, behavioral substitution with a sensory device (Fix Bar), and structured digital support. The purpose of this research is to evaluate the efficacy and safety of the investigational VapeAway system, a multi-component behavioral and nicotine-reduction intervention, for promoting cessation of nicotine-containing e-cigarette use in motivated adults. The primary objective is to determine if the VapeAway program can achieve a Continuous Abstinence Rate (CAR) of at least 25% at 30 days post-intervention completion, a rate which will be statistically compared to the historical spontaneous cessation rate of approximately 7%. Secondary objectives include assessing reductions in biochemical nicotine exposure (cotinine), vaping frequency, withdrawal symptoms, and electronic cigarette dependence, as well as characterizing the safety and tolerability profile of the intervention.

Participants will be asked to follow the VapeAway system (filters, Fix Bar and timeout periods) as prescribed by the protocol for about 42 days. During this time, participants should keep track of vaping sessions throughout the trial.

DETAILED DESCRIPTION:
This is a Phase II, single-arm, open-label, multi-center, interventional trial designed to assess the efficacy and safety of the VapeAway system for vaping cessation.

The study will enroll approximately 70 adult participants who are daily users of nicotine-containing e-cigarettes and are motivated to quit.

All enrolled participants will receive the active VapeAway intervention, which consists of a 42-day (±21 days) core program utilizing progressive nicotine tapering filters, a behavioral substitution device (Fix Bar), and a digital support system. The total study duration per participant will be approximately 90 days. The primary efficacy endpoint, the Continuous Abstinence Rate (CAR) at 30 days post-intervention completion, will be statistically compared to a predefined historical control spontaneous cessation rate of 7%.

The study will enroll adult males and females, aged 21 years and older, who are daily or near-daily users of nicotine-containing e-cigarettes for at least 3 months, have a saliva cotinine level ≥10 ng/mL, and score ≥4 on the Penn State Electronic Cigarette Dependence Index (PSECDI). Participants must be highly motivated to quit, as confirmed by standardized assessments (Likert scale, Motivation To Stop Scale, and the Preparation stage of the Transtheoretical Model).

The study includes several componenets:

1. Nicotine Tapering Filters: Participants will self-administer by attaching a new, study-supplied filter to their personal e-cigarette device each morning. Filters are used for all vaping sessions throughout the day and discarded after 24 hours. Participants will progress through the three filter levels (25%, 50%, 75% reduction) at scheduled intervals as follows:

   • Level 1 Filter (Days 1-14 ±7 days): Reduces nicotine delivery by 25% relative to baseline vaping device.

   • Level 2 Filter (Days 14-28 ±7 days): Reduces nicotine delivery by 50%.

   • Level 3 Filter (Days 28-42 ±7 days): Reduces nicotine delivery by 75%. Fix Bar: The Fix Bar is a behavioral substitution tool used in conjunction with nicotine tapering to replace the act of vaping. It can be used whenever the participant is vaping less than their baseline level, and it increases in use proportionally across each level.
   * Each Fix Bar contains three toothpicks and is refilled daily.
   * There are three distinct Fix Bars, one for each level of the program.
   * Participants will be assessed for their baseline vaping use calculated as hours per/day and will be instructed to increase Fix Bar usage (as a vaping replacement) for each timeout level, with target time replacements as follows:

   Level 1 (Days 1-14 ±7 days):
   * Week 1: Replace 15-20% of vaping time with Fix Bar
   * Week 2: Replace 30-35% of vaping time with Fix Bar

   Level 2 (Days 14-28 ±7 days):
   * Week 3: Replace 45-50% of vaping time with Fix Bar
   * Week 4: Replace 60--65% of vaping time with Fix Bar

   Level 3 (Days 28-42 ±7 days):
   * Week 5: Replace 80-85% of vaping time with Fix Bar
   * Week 6: Replace 95-100% of vaping time with Fix Bar
2. Use of the Fix Bar to replace vaping as oral fixation is optional however, the timeout periods are mandatory and will be tracked weekly. All participants will receive comprehensive training on the correct use of all system components at the Day 1 visit. Adherence will be monitored through weekly logs and reviewed at each study visit. Biochemical verification (saliva cotinine) will be performed at scheduled timepoints.
3. Digital Support System: Participant Support Messaging Protocol. As part of the intervention strategy for this study, all enrolled participants will receive ongoing motivational and supportive communication throughout the trial period and for a follow-up duration of up to 3 months post-intervention completion. The purpose of these communications is to enhance engagement, provide encouragement, and support participants in their efforts to reduce or cease vaping.
4. Text Message Support: Participants will receive up to five pre-written support text messages per week. These messages will be:

   * Designed to be motivational, encouraging, and engaging.
   * Focused on reinforcing positive behavior change, promoting well-being, and addressing common challenges in vaping cessation.
   * Tailored where possible to the participant's stage in the cessation journey.
5. Daily Text Messages: Separate from the support messages, participants will receive daily text messages reminding them of the number of timeout hours they are required to do for the day.

Upon completion of the intervention, participants will be followed for 30 days and a saliva cotinine test will be performed at the end of the follow-up period to confirm cessation.

ELIGIBILITY:
Inclusion Criteria:

* Age: Adults aged 21 years and older
* Current Vaping Behavior: Daily or near-daily use (≥5 days/week or at least 20 days per month) of nicotine-containing e-cigarettes for at least the past 3 months.
* Motivation and desire to quit as determined by all of the following three assessment tools:

  * Score of 4 or 5 on all 5-point Likert-type scale questions (see appendix)
  * Score of 6 or 7 on Motivation To Stop Scale (MTSS) (see appendix)
  * Participants must be classified in the Preparation stage of the Transtheoretical Model of behavior change (see appendix)
* Saliva Cotinine level ≥ 10 ng/ml
* Penn State Electronic Cigarette Dependence Index (PSECDI) of at least 4 and above
* Willingness to participate in the study and all study requirements
* Willingness to not use any other nicotine-containing products for the duration of the study
* Ability to attend visits and provide informed consent

Exclusion Criteria:

* Mental Health Concerns with a score above the following thresholds:

  * PHQ-2 score ≥ 2 (see appendix)
  * GAD-2 score ≥ 2 (see appendix)
* Use of Other Tobacco or Nicotine Products:

  * Use of any nicotine products except for vaping, including combustible tobacco (e.g., cigarettes) or other non-e-cigarette nicotine delivery systems within the past 30-days
* Current Substance or alcohol Use Disorder:

  * Self-reported or medically diagnosed substance use disorder (excluding nicotine), unless in sustained remission (>12 months).
  * Illicit drug use in the past 60 days
  * Screening positive for alcohol use disorder in past year
* Medical Contraindications:

  * Any serious medical condition or medication that would contraindicate participation in a behavioral cessation trial (to be defined and assessed by study physician or PI).
  * Pregnant or breastfeeding
  * Symptomatic cardiovascular disease
  * Participation in another smoking/vaping cessation trial

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-12-24 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Vaping Cessation | up to 90 days
  To determine the prevalence of vaping abstinence (quit rates) with the VapeAway system at 30 days after completion of the program (intervention period) verified by self-reporting and biochemical testing

SECONDARY OUTCOMES:
Filter Compliance | Up to 63 days
  Percent of time the subject vaped with use of filter

CONTACTS AND LOCATIONS:
Overall Officials: Mendel Goldfinger, MD, Principal Investigator — VapeAway
Locations (1):
- Prime Infusion, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No